CLINICAL TRIAL: NCT03348943
Title: Comparative Analysis of Motor Performance in People With Cerebral Palsy (Spastic Hemiparesis) by Virtual Task.
Brief Title: Motor Learning in People With Cerebral Palsy by Using Virtual Reality.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carlos Bandeira de Mello Monteiro, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 61384416.3.0000.8028
Record Dates: First submitted 2017-06-01; First posted 2017-11-21 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Right hemiparesis, right upper limb (Active Comparator): Individuals with right hemiparesis Cerebral Palsy that will perform the tasks with the affected upper limb.
  Interventions: Behavioral: Right hemiparesis, right upper limb.
- Right hemiparesis, left upper limb (Experimental): Individuals with right hemiparesis Cerebral Palsy that will perform the tasks with the non-affected upper limb.
  Interventions: Behavioral: Right hemiparesis, left upper limb
- Left hemiparesis, left upper limb (Active Comparator): Individuals with left hemiparesis Cerebral Palsy that will perform the tasks with the affected upper limb.
  Interventions: Behavioral: Left hemiparesis, left upper limb
- Left hemiparesis, right upper limb (Experimental): Individuals with left hemiparesis Cerebral Palsy that will perform the tasks with the non-affected upper limb.
  Interventions: Behavioral: Left hemiparesis, right upper limb

INTERVENTIONS:
Behavioral: Right hemiparesis, right upper limb. — Individuals with right hemiparesis Cerebral Palsy that will perform the tasks with the affected upper limb.
  Arms: Right hemiparesis, right upper limb
Behavioral: Right hemiparesis, left upper limb — Individuals with right hemiparesis Cerebral Palsy that will perform the tasks with the non-affected upper limb.
  Arms: Right hemiparesis, left upper limb
Behavioral: Left hemiparesis, left upper limb — Individuals with left hemiparesis Cerebral Palsy that will perform the tasks with the affected upper limb.
  Arms: Left hemiparesis, left upper limb
Behavioral: Left hemiparesis, right upper limb — Individuals with left hemiparesis Cerebral Palsy that will perform the tasks with the non-affected upper limb.
  Arms: Left hemiparesis, right upper limb

SUMMARY:
Cerebral Palsy (CP) is a group of permanent disorders that affect movement and posture due to a non-progressive lesion in the immature brain occurring in fetal brain development or in infancy. These disorders are often associated with changes in sensation, learning, body perception, communication and behavior. People with CP present variable difficulties in muscle action. With increasing access to computer-aided accessibility, rehabilitation programs have increasingly used virtual reality (VR) environments to provide functional tasks. Virtual reality research in individuals with cerebral palsy has demonstrated improvements in gross motor functions and functional disabilities in mobility, and is a good device for rehabilitation. The present research is a cross-sectional study. For this study 40 individuals aged over six years (with task comprehension) of both gender who have a clinical diagnosis of spastic hemiparetic Cerebral Palsy will be evaluated. Thus, the present study aims to compare the motor function of the committed and uncommitted body side by performing tasks in virtual reality.

DETAILED DESCRIPTION:
METHOD The present research is a cross-sectional study. The study will be carried out at the School of Special Education Don Bosco, Rio Branco, Acre.

PARTICIPANTS (CASE) For this study 40 individuals aged over six years (with task comprehension) of both gender who have a clinical diagnosis of spastic hemiparetic Cerebral Palsy will be evaluated.

STUDY DESIGN The individuals selected will be divided according to the affected body side, forming a first group categorized by RH (Right Hemiparetic) and a second LH (Left Hemiparetic), and for the accomplishment of the activity in the RH group half will start the task with the affected side and than with the unaffected side and the same will be reproduced in the LH group. Before performing the matching Timing task, individuals will perform a simple reaction time (RT) task, with 14 repetitions in each task.

Next, they will perform 20 attempts of the Timing task in the acquisition phase (0.5 second speed between the firings of each sphere - level 4), after 10 minutes without contact with the task the subjects will carry out 5 attempts for the Retention phase at the same speed as the acquisition phase. Then the subjects will perform 5 more attempts for the transfer phase with change in the speed of the task (0.25 seconds between the firings of each sphere - level 5). After the task is finished, the TR will be applied again.

INSTRUMENTS Timing Software Coincident For the data collection will be used a software of games created in partnership with the group of Information Systems of the School of Arts, Sciences and Humanities, EACH-USP. The game proposes a Coincident Timing task, which displays on the computer screen 10 spheres that light up (red light) in sequence until reaching the last ball that is considered the target (Green light). The participant can have immediate feedback of correctness or error of the task through different sounds (Auditory Interaction) and through visual images (Visual Interaction) that change color previously demonstrated to them.

Software TRT_S (Simple Reaction Time) Other software used was TRT_S2012. Which was constructed and validated by Crocetta et al. The software proposes a simple TRT test consisting of the appearance of a yellow square (parameterizable) in the center of the monitor at predefined time intervals (ranging from 1.5 to 6.5 ms - these intervals were identical in both Software) and, when the stimulus is applied, the participant should react as quickly as possible by pressing the spacebar on the computer keyboard.

Procedure and design Participants will perform the task individually in a quiet room, with only the experimenter, who will provide the instructions. The computer monitor will be positioned on a desk. Participants will remain seated in the chair with height adjusted according to the needs of each. In addition, a footrest will be available if needed. The functional assessment scales will be performed at the beginning of the research, the experimenter will explain the task verbally and perform a demonstration of the game's functioning and interfaces (Kinect for Windows®, touch the computer key or touchscreen).

ELIGIBILITY:
Inclusion Criteria:

* classification of gross motor function with levels I and II according to the Gross Motor Function Classification System (GMFCS),
* MACS (Manual Ability Classification System) classification between levels I and II.

Exclusion Criteria:

* over 20 years;
* comorbidities that prevent the accomplishment of the activity;
* people with significant visual and cognitive impairment;
* those who have undergone chemical blockade or upper limb surgery for less than six months

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Difference in performance of the Coincident Timing task between participants with right hemiparesis and participants with left hemiparesis | 6 months.
  There will be differences between right and left hemiparesis regarding coincident timing (e.g. patients with left hemiparesis will have a worse time in milliseconds that patients with right hemiparesis).

CONTACTS AND LOCATIONS:
Overall Officials: Carlos BM Monteiro, Ph.D., Principal Investigator — University of Sao Paulo
Locations (1):
- Escola de Artes,Ciencias e Humanidades da Universidade d Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided